CLINICAL TRIAL: NCT05653570
Title: Electrical Stimulation for Erector Spinae Plane Catheter Insertion: A Randomized Controlled Trial
Brief Title: Electrical Stimulation for Erector Spinae Plane Catheter Insertion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jan Boublik, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 68478
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2025-04-21 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain, Acute; Shoulder Pain
Keywords: erector spinae plane; electrical stimulation
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ultrasound Guidance Only (Active Comparator)
  Interventions: Diagnostic Test: Ultrasound
- Electrical stimulation and Ultrasound Guidance (Experimental)
  Interventions: Diagnostic Test: Electrical stimulation; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Electrical stimulation — Electrical stimulation will be used to confirm needle and catheter placement within the interfascial plane between the erector spinae muscle and thoracic transverse process.
  Arms: Electrical stimulation and Ultrasound Guidance
Diagnostic Test: Ultrasound — Ultrasound guidance will be used to visualize needle and catheter placement within the interfascial plane between the erector spinae muscle and thoracic transverse process.

SUMMARY:
The erector spinae plane (ESP) block has been studied for analgesia in shoulder surgery as a phrenic nerve-sparing alternative. However, successful ESP catheter placement appears multifactorial, with failure mechanisms including lamination, plane collapse, or catheter overcoiling. Electrical stimulation (ES) is a common technique used in regional anesthesia to detect possible intraneural placement. ES of the erector spinae muscle complex may objectively guide proper interfascial catheter placement and improve local anesthetic spread. The primary goal of this study is to establish if ESP catheter placement with the addition of ES to ultrasound (US) guidance facilitates accurate catheter placement. This study will further characterize postoperative analgesia and the incidence of brachial plexus stimulation for patients who receive ES-assisted ESP catheter placement.

ELIGIBILITY:
Inclusion Criteria:

* elective total or total reverse shoulder arthroplasty

Exclusion Criteria:

* inability to provide consent
* history of active opioid use
* emergency procedures
* shoulder arthroscopy
* partial shoulder replacement
* shoulder resurfacing
* any revision shoulder surgery
* any indwelling deep brain stimulator, pacemaker, and/or other neurostimulators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with erector spinae muscle stimulation via stimulating catheter | Immediately after catheter placement (up to 5 minutes to assess)
  Successful erector spinae plane needle and catheter insertion means that the needle/catheter is deep to the myofascia of the erector spinae muscle complex and superficial to the intertransverse ligaments / transverse process. Thus, any stimulation of the catheter after its placement in the erector spinae muscle complex seen under ultrasound or perceived by the patient will be documented as catheter placement failure. No visualized or perceived stimulation of the erector spinae muscle complex will be documented as catheter placement success.

SECONDARY OUTCOMES:
Time to perform erector spinae plane catheter | During catheter placement (up to 20 minutes)
  Time for catheter placement will begin when the US probe first touches the patient and end when the inner stimulating catheter hub meets the skin. If no visual identification of the target erector spinae plane (US) and no evoked motor respoinse (US+ES) is achieved within 10 minutes, the placement will be considered a failure, and the primary end point will be recorded as 10 minutes. If a catheter cannot be placed per protocol within 20 minutes, the placement will be considered a failure, and the primary endpoint will be recorded as 20 minutes. In such cases, the subject will have a catheter placement attempt using the alternative method. Subjects who do not have a catheter placed as per their randomized group protocol will be removed from further study.
Worst pain score ratings in the postanesthesia care unit (PACU) | as soon as patient can respond in PACU (up to 1 hour)
  As soon as the patient is able to respond verbally in the PACU, the subject will be asked to rate their pain on an 11-point numeric rating scale (NRS, 0 being no pain and 10 being worst possible pain)
Highest and lowest vertebral level of sensory change after local anesthetic bolus | preoperatively, 30 minutes after local anesthetic bolus
  We will administer cold spray (name, manufacturer location) 3 cm lateral to the spinous process from C1 to T12, and document the highest and lowest dermatomal levels of when the patient detects a difference in temperature sensation compared to the contralateral side.
Incidence of brachial plexus or intercostal stimulation via stimulating catheter before local anesthetic bolus | preoperatively, prior to local anesthetic bolus (up to 5 minutes)
  Prior to local anesthetic bolus, any perceived stimulation of an intercostal muscle or in the distribution of the brachial plexus on the operative side, including but not limited to twitching of or warmth of skin overlying the deltoid, biceps, triceps, supraspinatus, infraspinatus, pectoralis major/minor, and teres major/minor, will be documented.
Incidence of brachial plexus or intercostal stimulation via stimulating catheter after local anesthetic bolus | preoperatively, 30 minutes after local anesthetic bolus
  30 minutes after local anesthetic bolus, any perceived stimulation of an intercostal muscle or in the distribution of the brachial plexus on the operative side, including but not limited to twitching of or warmth of skin overlying the deltoid, biceps, triceps, supraspinatus, infraspinatus, pectoralis major/minor, and teres major/minor, will be documented.
Opioid consumption in the PACU | from admission to discharge from the PACU (average approximately 2 hours)
  The subject's total opioid administration in the PACU will be documented and converted to oral morphine milliequivalents (MME).
Opioid consumption on postoperative day (POD) 1 | POD1 (24 hours)
  The subject's total opioid administration on POD1 will be documented and converted to oral morphine milliequivalents (MME).
Opioid consumption on postoperative day (POD) 2 | POD2 (24 hours)
  The subject's total opioid administration on POD2 will be documented and converted to oral morphine milliequivalents (MME).
Opioid consumption on postoperative day (POD) 3 | POD3 (24 hours)
  The subject's total opioid administration on POD3 will be documented and converted to oral morphine milliequivalents (MME).
Average postoperative pain on postoperative day (POD) 1 | POD1 (24 hours)
  The subject's average postoperative pain score ratings will be calculated on POD 1. Pain scored on an 11-point numeric rating scale (NRS, 0 being no pain and 10 being worst possible pain)
Average postoperative pain on postoperative day (POD) 2 | POD2 (24 hours)
  The subject's average postoperative pain score ratings will be calculated on POD 2 Pain scored on an 11-point numeric rating scale (NRS, 0 being no pain and 10 being worst possible pain)
Average postoperative pain on postoperative day (POD) 3 | POD3 (24 hours)
  The subject's average postoperative pain score ratings will be calculated on POD 3 Pain scored on an 11-point numeric rating scale (NRS, 0 being no pain and 10 being worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Boublik, MD, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No